CLINICAL TRIAL: NCT06281392
Title: Effect of an Artificial Intelligence System on the Detection of Dysplasia During Colonoscopy in Patients With Long-standing Inflammatory Bowel Disease: a Randomized Study (EIIDISIA Study)
Brief Title: Artificial Intelligence and Dysplasia Detection in Inflammatory Bowel Disease (EIIDISIA Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Antonio López-Serrano, Chief of Endoscopy Section, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: CEIm: 106/23
Record Dates: First submitted 2023-11-27; First posted 2024-02-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Diseases; Dysplasia
Keywords: Inflammatory Bowel Disease; Virtual chromoendoscopy; NBI; CADe; Dysplasia
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colonoscopy assisted by CADe (Experimental)
  Interventions: Device: CADe system
- Virtual Colonoscopy with NBI (Active Comparator)
  Interventions: Device: NBI

INTERVENTIONS:
Device: CADe system — Colonoscopy assisted by an artificial intelligence system (CADe).
  Arms: Colonoscopy assisted by CADe
Device: NBI — Virtual colonoscopy assisted by NBI
  Arms: Virtual Colonoscopy with NBI

SUMMARY:
Randomized clinical study analyzing the efficacy of colonoscopy assisted by the Computer Aided Detection (CADe) system compared to virtual chromoendoscopy with Narrow Band Imaging (NBI) in the detection of colon dysplasia in patients with long-standing inflammatory bowel disease (IBD).

ELIGIBILITY:
INCLUSION CRITERIA:

* Adults (age ≥18 years).
* Patients with IBD meeting the following criteria:
* Diagnosis of IBD confirmed by clinical and histological evidence.
* Disease extent (Montreal classification): 1) For Ulcerative Colitis (UC), Extensive colitis (E3): involvement proximal to the splenic flexure; or, Left-sided colitis (E2): involvement distal to the splenic flexure. 2) For Crohn's Disease (CD): Colon-only involvement (L2); or, Ileocolonic involvement (L3).
* Disease duration > 7 years.
* Patients with concommitant Primary Sclerosing Cholangitis, regardless of the extent of colonic involvement and disease duration.
* Written consent from the patient to undergo colonoscopy (signed informed consent).

EXCLUSION CRITERIA:

* Personal history of colorectal cancer (CRC).
* Previous colectomy (partial or complete).
* Coagulopathy preventing biopsy or polypectomy/mucosal resection.
* Colonoscopy performed in the last 6 months.
* Pregnant or lactating women.
* Ulcerative colitis with involvement limited to the rectum or Proctitis (Montreal E1).
* Inadequate colonic preparation due to uncleavable fecal residue during colonoscopy: Boston Bowel Preparation Scale (BBPS) = 0 or 1 in any colon segment.
* Presence of inflammatory activity due to IBD on endoscopy:1) For UC: Endoscopic Mayo Score ≥ 2. 2) For CD: Simplified Endoscopic Activity Score (SES-CD) > 5.
* Incomplete lower digestive endoscopy (failure to reach the cecum).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
"Per lesion" dysplasia detection rate (DDR) | Immediately after the procedure
  Proportion of dysplastic lesions in relation to all the lesions analyzed that were detected by Artificial Intelligence System (CADe) or Virtual chromoendoscopy with NBI in patients with long-standing Inflammatory bowel disease who undergo surveillance colonoscopy
"Per patient" dysplasia detection rate (DDR) | Immediately after the procedure
  Proportion of patients with dysplastic lesions in relation to all the patients with long-standing Inflammatory bowel disease included in the study detected by Artificial Intelligence System (CADe) or Virtual chromoendoscopy with NBI

SECONDARY OUTCOMES:
Duration of endoscopic examination | Immediately after the procedure
  Median (IQR) examination time (in minutes) (including total, insertion, and withdrawal time) required by Artificial Intelligence System (CADe) or Virtual chromoendoscopy with NBI

CONTACTS AND LOCATIONS:
Overall Officials: Antonio López-Serrano, PhD, Principal Investigator — Hospital Universitari Dr. Peset, Valencia (Spain)
Locations (1):
- Antonio López-Serrano, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No